CLINICAL TRIAL: NCT06706648
Title: Examining the Role of Nursing-Led Psychological Capital Interventions on Staff Nurses' Occupational Hardiness and Engagement: a Randomized Controlled Trial
Brief Title: Examining the Role of Nursing-Led Psychological Capital Interventions on Staff Nurses' Occupational Hardiness and Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Alaa El Din Moustafa Hamed Abd Elaleem, Lecturer of Psychiatric and mental health Nursing, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUNURREC2024340/13
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-05

CONDITIONS: Occupational Hardiness; Work Engagement; Psychological Capital Interventions
Keywords: Nurses; Occupational Hardiness; Work Engagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention)
- Study Group (Experimental): Study group who recived Nursing-Led Psychological Capital Interventions
  Interventions: Behavioral: Nursing-Led Psychological Capital Interventions

INTERVENTIONS:
Behavioral: Nursing-Led Psychological Capital Interventions — The participating nurses received session about Nursing-Led Psychological Capital Interventions
  Arms: Study Group

SUMMARY:
This study aimed to evaluate the effect of nursing-led psychological capital intervention on nurses' occupational hardiness and work engagement. The main hypothesis was that staff nurses who received tailored nursing-led psychological capital intervention (study group (SG)) will demonstrate significantly greater improvements in occupational hardiness and work engagement compared to those who received an educational booklet (control group (CG)).

DETAILED DESCRIPTION:
This study recruited nurses working 12 hours per shift for 144-180 hours a month at Damietta university hospitals in Damietta Governorate, Egypt. Nurses who were licensed staff nurses, worked in ICU, and had at least 6 months of experience been included in the analysis. In contrast, nurses who were involved in any other intervention program within the last 12 months, working in either wards or any department rather than ICU, or holding an administrative position were excluded. The psychological capital intervention program was developed based on the principles of psychological capital, which include hope, optimism, resilience, and self-efficacy. The intervention aimed to train participants in enhancing their psychological resources. This included fostering hope and optimism, building resilience to cope with challenges, and strengthening self-efficacy to manage job demands. The intervention assists staff nurses in cultivating a positive mindset, boosting their work engagement, and adapting to challenges in the workplace. Ultimately, it sought to enhance their occupational hardiness, foster a greater sense of work passion, and strengthen their career commitment.

Prior to the implementation of the PCI program, interviews were held with potential participants and nursing managers. These interviews explored staff nurses' perceptions of what constitutes good performance, the barriers they face in achieving it, the factors that support them in providing high-quality care, the tasks which they perceive as challenging, and the reasons which make them avoid these challenges. The discussions also focused on factors influencing occupational hardiness and work engagement, including nurses' ability to adapt to new challenges, their work passion, and career commitment. This comprehensive understanding of the work environment was used to design a tailored Psychological Capital Intervention (PCI) program, incorporating customized examples to address these specific challenges, with the goal of enhancing both occupational hardiness and work engagement among staff nurses.

Committee included Five-expert in nursing field as the following one nursing administration professor, one chief of nursing officer (CNO), Deputy of CNO for critical area, Critical area nursing supervisor and one staff nurse with master's degrees were asked for suggestions on the content and structure of the intervention materials. The intervention materials were modified based on their suggestions and sent back to the committee for approval. Then the intervention materials were pilot tested to ensure their quality and clarity.

ELIGIBILITY:
Inclusion Criteria:

* ICU Nurse Nurse hold license. More than 6 Months of Experience Aged Between 20-60

Exclusion Criteria:

Working in any place rather than ICU. attended training about psychological capital intervention in the last 12 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Occupational hardiness | 3 months
  Occupational hardiness is measured by Occupational hardiness questionnaire (OHQ) was developed by Moreno-Jiménez and colleagues, (2014). This questionnaire is used to measure hardihood and resoluteness among employees. It is a 5-point Likert- scale with 17 items and responses range from 1 = Strongly Disagree to 5 = Strongly Agree. This scale assessed the influence of the three aspects of employees' hardiness, namely, commitment, control, and challenge. Sample items on the OHQ are: "I do everything I can to make sure I control the results of my work" and "In my job I feel attracted to tasks and situations involving a personal challenge". Cronbach's alpha reliability coefficients for the three sub-scales of this scale as reported by the developers were.78, .73, and 0.72 respectively for commitment, control, and challenge. Cronbach's alpha for the scale as a whole was .75, indicating strong internal consistency reliability.

SECONDARY OUTCOMES:
Work Engagement | 3 months
  Work Engagement is measured by Work Engagement Scale (WES-17) was developed by Schaufeli and Bakker, (2006). This scale to measure three related factors of work engagement: vigour, dedication, and absorption. Categorized by levels of high energy and mental resilience. It consists of 17 items divided into three domains and as follows vigor represented 6 items. vigour describes a willingness to persevere in the face of obstacles in the workplace or the willingness to continue to invest effort in one's work when confronted with a challenge. Dedication represents 5 items, it implies heavy involvement in one's work and through this work, one experiences a sense of challenge, pride, and inspiration, Individuals with high levels of dedication see their work as meaningful and inspiring. Lastly Absorption represented 6 items, it is defined as being happily engrossed in and concentrated on one's work, where time seems to pass rather quickly, and where one has difficulty detaching themselves.

CONTACTS AND LOCATIONS:
Locations (1):
- Damietta University, Damietta, Damietta Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No